CLINICAL TRIAL: NCT05671055
Title: CogMS - A Real-world Study Into Cognitive Impairment in People With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: icometrix (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: ICO-S-001
Record Dates: First submitted 2022-11-28; First posted 2023-01-04 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Multiple Sclerosis
Keywords: Cognition
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Main arm: Use of icompanion through will all assessments are performed
  Interventions: Other: Custom study version of icompanion app

INTERVENTIONS:
Other: Custom study version of icompanion app — Patients complete patient-reported outcomes on cognition and covariates, as well as objective cognitive tests through a version of icompanion app customized specifically for this study. Patients complete all assessments remotely in an at-home situation.

SUMMARY:
The present study will investigate the correlation between objective and subjective cognition in multiple sclerosis. The study will also investigate the impact of covariates such as fatigue and depression, the relationship with the Expanded Disability Status Scale (EDSS) and brain volumetrics as measured on magnetic resonance imaging (MRI). Additionally, the study will provide insights into patients' experiences with cognition, and the usability of the used objective cognitive assessments.

DETAILED DESCRIPTION:
Cognitive impairment is a significant burden that affects 43 to 70% of persons with multiple sclerosis (pwMS) 1. Cognitive problems have been observed in the earliest stages of multiple sclerosis (MS) and multiple studies have provided evidence for the predictive value of early cognitive impairment for future disease progression 2-6. However, cognitive function is not often discussed with pwMS or routinely assessed by healthcare providers (HCPs) leading to sub-optimal treatment of cognitive problems in MS 7. Furthermore, cognitive dysfunction that can be reliably detected by objective measures is poorly recognized by pwMS, resulting in a disconnect between objective and subjective measures of cognitive function 8-10.

The present study will investigate the correlation between what cognitive problems people with MS perceive and what objective cognitive testing actually shows. This study will also provide insights about the presence of this disconnect in different strata of the Expanded Disability Status Scale (EDSS) 11, and the relationship with possible confounders (MS symptoms, fatigue, etc.) and brain volumetrics as measured on magnetic resonance imaging (MRI).

Study Design:

CogMS is an observational, cross-sectional, remote, real-world study of cognitive function in patients with multiple sclerosis. We will investigate the correlation between subjective and objective patient self-evaluations of cognitive function while also investigating the prevalence of objective cognitive impairment in different EDSS strata of pwMS. MS patients will be stratified by EDSS to evaluate the correlation between objective and subjective cognition in three different EDSS strata (EDSS 0 - 2; 2.5 - 3.5; 4.0 - 5.5) and the occurrence of objective cognitive dysfunction in these EDSS stages of MS.

All data will be captured using the icompanion app in a remote, non-clinical setting (i.e., patient's home) within three weeks of patient onboarding. In the icompanion app, patients will be asked to perform the icognition cognitive test battery together with patient-reported outcomes (PROs) for subjective cognition, MS symptoms, prEDSS, depression and fatigue. If available, a recent (max. 6 months) MRI scan will be provided from which volumetric measurements can be calculated using icometrix' icobrain software.

Finally, patients will be asked to answer questions on their experiences with cognition since diagnosis, their preferences and opinions about cognition as a treatment goal, and the usability of the icognition battery, and the preference compared to paper-based neuropsychological tests.

ELIGIBILITY:
Inclusion Criteria:

* Providing a signed informed consent
* Aged between 18 and 65 years old
* MS diagnosis (CIS, RRMS)
* Absence of hand function problems which limit the use of a device like a smartphone
* No history of relapse with onset 30 days prior to start of study
* No other major neurological or psychiatric disorders
* No history of cognitive rehabilitation treatment

Exclusion Criteria:

* Disease duration longer than 15 years
* Patients with established cognitive disorders other than MS
* Drug and/or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 300 CIS/RRMS patients, aged 18 to 65 (inclusive), with a maximum disease duration of 15 years.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2023-01-07 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Neuro-QoL cognitive | Single cross-sectional time-point (max 2 months after signing ICF)
  The Neuro-QoL (Quality of Life in Neurological Disorders) is a patient-reported outcome for subjective cognitive problems Minimum and maximum values: 8-40 (t-score: 17.3-64.2). High scores indicate better (desirable) self-reported health.
icognition Symbol test score | Single cross-sectional time-point (max 2 months after signing ICF)
  The icognition Symbol test is a smartphone-based symbol substitution test for information processing speed Minimum and maximum values: to be determined by a separate study which is being finalised High scores indicate better (desirable) self-reported health.
icognition Dot test score | Single cross-sectional time-point (max 2 months after signing ICF)
  The icognition Dot test score is a smartphone-based test for visual working memory Minimum and maximum values: to be determined by a separate study which is being finalised High scores indicate better (desirable) self-reported health.
icognition Digit test score | Single cross-sectional time-point (max 2 months after signing ICF)
  The icognition Digit test score is a smartphone-based test for working memory Minimum and maximum values: to be determined by a separate study which is being finalised High scores indicate better (desirable) self-reported health.

SECONDARY OUTCOMES:
prEDSS | Single cross-sectional time-point (max 2 months after signing ICF)
  is a patient-reported outcome (PRO) version of the Expanded Disability Status Scale (EDSS), the current golden standard method for assessing disability (progression) in MS.
  Minimum and maximum values: 0-10 Low scores indicate better (desirable) self-reported health.
Neuro-QoL fatigue | Single cross-sectional time-point (max 2 months after signing ICF)
  Neuro-QoL Fatigue is a patient-reported outcome for fatigue Minimum and maximum values: 8-40 (t-score: 29.5-74.1). Low scores indicate better (desirable) self-reported health.
Beck's depression inventory | Single cross-sectional time-point (max 2 months after signing ICF)
  The BDI is a 21-question multiple-choice self-report psychometric tests for measuring the severity of depression.
  Minimum and maximum values: 0-63. Low scores indicate better (desirable) self-reported health.
MRI volumetric variables | at time of enrolment in study (in case MRI of <6months is available)
  icobrain volumetric MRI measurements: whole brain volume and atrophy, grey matter volume and atrophy, lesion load, total lesion volume, volume of new lesions, volume of enlarging lesions, volume of shrinking lesions, lesion volume and volume changes assessed locally (i.e. juxtacortical, periventricular, deep white matter, infratentorial)
System usability score (cognitive smartphone-based tests) | Single cross-sectional time-point (max 2 months after signing ICF)
  Usability questionnaire
Preference icognition vs. paper-based assessments | Single cross-sectional time-point (max 2 months after signing ICF)
  Likert scale [0-5]
SymptoMScreen | Single cross-sectional time-point (max 2 months after signing ICF)
  Questionnaire assessing the severity of the twelve most common MS Symptoms Minimum and maximum values: 0-6 Low scores indicate better (desirable) self-reported health.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Nagels, Prof., Principal Investigator — UZ Brussel - icometrix
Locations (10):
- United States (5):
  - UCHealth, Aurora, Colorado
  - Brain Health Center of the Rockies, Fort Collins, Colorado
  - Dent Neurologic Institute, Buffalo, New York
  - The Boster Center for Multiple Sclerosis, Columbus, Ohio
  - Texas Neurology, Dallas, Texas
- Belgium (4):
  - GZA Antwerpen, Antwerp
  - Imelda Ziekenhuis, Bonheiden
  - AZ Sint-Jan Brugge, Bruges
  - UZ Brussel, Jette
- University of Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No